CLINICAL TRIAL: NCT03319095
Title: Intravaginal Electrical Nerve Stimulation to Achieve a Voluntary Contraction in Women With Non-contracting Pelvic Floor: a Randomized Controlled Trial
Brief Title: Intravaginal Electrical Nerve Stimulation in Women With Non-contracting Pelvic Floor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Flávia Ignácio Antônio Vassimon, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 73055317.8.0000.5440
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Pelvic Floor; Muscle; Contraction; Electric Stimulation Therapy
Keywords: pelvic floor, muscle, electrical stimulation, physiotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The main investigators and assessor will be blinded in relation to the allocation of participants in the groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control group: participants will receive only verbal instructions on PFM anatomy and function during the first assessment when women will be required to contract their pelvic floor muscle. The participants will have no contact with the service until the second assessment
- Intervention (Active Comparator): Intravaginal Electrical Nerve Stimulation: participants will be submitted to Intravaginal Electrical Nerve Stimulation
  Interventions: Device: Intravaginal Electrical Nerve Stimulation

INTERVENTIONS:
Device: Intravaginal Electrical Nerve Stimulation — The Intervention group will receive Intravaginal Electrical Nerve Stimulation using Quark® Dualpex equipment, once per week during 8 weeks. The selected current will be biphasic, and the stimulation parameters will be: 50 Hz frequency, pulse width of 200 microseconds, contraction time (Ton) of 5 seconds, relaxation time (Toff) of 10 seconds, intensity of current defined according to the sensitivity (tolerance) of the patient, and total stimulation time of 20 minutes once a week delivered by an experienced Physiotherapist. In the last 10 minutes of each electrical nerve stimulation session women will be requested to perform voluntary PFM contractions along with the contractions induced by the electrical stimulation. Women will not be instructed to perform any aditional exercise or therapy at home.
  Arms: Intervention

SUMMARY:
It is estimated that about 30% of women cannot voluntarily contract the pelvic floor muscles (PFM). PFM training (PFMT) represents the first therapeutic option for the treatment of female urinary incontinence (UI), however the inability to contract this muscle makes PFMT unfeasible. The primary objective of this project is to evaluate clinically the efficacy of intravaginal electrical stimulation associated with verbal instructions to provide the ability of women to contract voluntary their PFM. The secondary objective is to evaluate the UI prevalence and impact on quality of life.

DETAILED DESCRIPTION:
This is a randomized controlled trial. A simple randomization procedure will be conducted using computer generated list. This list will be kept with a secretary not involved with the research. A concealed allocation will be performed. All participants will be recruited at Rehabilitation Center of the Clinical Hospital of Ribeirão Preto Medical School, University of São Paulo. The primary outcome of the study will be vaginal palpation, to differentiate women capable or not capable to perform a PFM contraction. The secondary outcome will be measured using the ICIQ- UI SF questionnaire.

To analyze the proportions of improvement after the intervention in relation to primary outcome we will consider the proportion of women with values equal or above 2 and 3 as specified in the outcome measure section, using the modified oxford grading scale. The sample size calculation will be done based in a pilot study after the study initiate (after registration) considering we found no data from a RCT investigating exactly the same intervention. The study of Vasconcelos et al. (2017) that investigated a similar intervention in the same population performed a sample size calculation using a test of differences between proportions and Fisher's exact test based in the proportion of change in the group receiving electrical stimulation ( 0.35 point) and in the control group (CG) (0.13 point). Considering a significance level of 5% and 80% test power, in the comparison between the intervention group (IG) and control group (CG), the minimum number indicated was 61 participants per group; however as the intervention was not exactly the same and the control group received instructions to perform home training we intend to do this calculation again based in a pilot sample after the study initiate (after registration).

As stated before in the initial registration, the sample size calculation was conducted based on a pilot test carried out by the researcher. The sample calculation was used for qualitative data (primary outcome measure) and non-paired sample based on the proportion of improvement after the intervention. The sample calculation compared n=14 in the control group and n= 9 in the intervention group. Considering the proportion of improvement, after intervention, in women with values equal or above 2 is suggested that a sample size of 14 participants per group would be adequate to see between group differences at power=0.90 and α=0.05. In a second situation, the proportion of improvement will be considered as a value equal or above 3, in this case a sample size of 28 participants per group would be adequate to see between group differences at power=0.80 and α=0.05, and 37 participants per group would be adequate to see between group differences at power=0.90 and α=0.05.

Data analysis The data will be analyzed initially through descriptive statistics, which will enable the characterization of the sample regarding the variables collected. This methodology has as basic objective to synthesize a series of values of the same nature, allowing a global view of the variation of these values, organizing and describing the data through tables of frequencies and descriptive measures.

To verify the association between the categorical variables, the data will be submitted to Fisher's exact test. The association quantification will be measured through logistic regression models, where the crude odds ratio with its respective 95% confidence intervals will be calculated.

The analysis of variance (ANOVA) will be used to verify the homogeneity between the groups of quantitative variables. The Student's t-test will be used to compare two means from unpaired samples. To test whether the variances of the two groups are statistically equal, and if the data follows the normal distribution, the PROC TEST procedure of the SAS software will be used. The mixed effects linear models (random and fixed effects) will be used for the analysis of the ICIQ-S questionnaire. This method is used in the analysis of data where the responses of the same individual are grouped and the assumption of independence between observations in the same group is not adequate (Schall, 1991). In the mixed-effects model used, individuals will be considered as random effects and, as fixed effects, the groups, the times and the interaction between them. The adjustment of the model will be done through the PROC MIXED procedure of the statistical software SAS.

The results will be reported as estimates of effect size. In relation to the primary outcome we will present the proportion of improvement, crude odds ratio with respective confidence intervals of 95%. For the secondary outcome measure we will present mean difference and 95% CI).

Data will be analyzed Independent of compliance to intervention (intention to treat analysis). A secondary per-protocol analysis will be done to verify the effect of trial adherence on the primary outcome. This analysis will include only women who received at least 80% of the physiotherapy sessions.

A sensitivity analysis will be performed if necessary to adjust for possible baseline imbalances.

All statistical analyzes will be performed using the SAS® 9 statistical software. The level of significance adopted for all tests will be 5%.

Quality assurance plan that addresses data validation and registry procedures, including any plans for site monitoring and auditing.

Data checks to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.

Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources (for example, medical records, paper or electronic case report forms, or interactive voice response systems).

Data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information if used (for example, World Health Organization Drug Dictionary, MedDRA), and normal ranges if relevant.

Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management.

.

ELIGIBILITY:
Inclusion Criteria:

* Women who are routinely referred to the Lucy Montoro Rehabilitation Center of the Hospital das Clínicas of the University of São Paulo at Ribeirão Preto Medical School - HCFMRP-USP for the physiotherapeutic treatment of pelvic floor dysfunctions;
* Pelvic floor muscle function grade 0 (zero) or 1 evaluated by bidigital palpation (Modified Oxford Scale);
* Consent to participate in the study and signing of the free and informed consent form.

Exclusion Criteria:

* Women with associated neurological pathologies;
* Symptoms of vaginal or urinary tract infection;
* Prolapses classified above grade 2;
* Suspected or confirmed pregnancy and cognitive deficit that compromises the procedure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Bidigital Vaginal Palpation | 30 minutes
  The primary outcome will be assessed by bidigital vaginal palpation using the modified Oxford scale at baseline and after 10 weeks. The correct contraction of the PFM will be considered as the action of occlusion and elevation of the PFM around the examiner's fingers in the ventral and cranial directions. Therefore, it will be considered a clinically relevant improvement to obtain a score above 3 on the modified Oxford scale.
  The examination will be performed following the following steps:
  * The participant will receive information about the procedure, and basic anatomy of the PFM.
  * She will be placed in dorsal decubitus, with hips and knees flexed, feet supported and legs apart;
  * The examiner using a procedure glove will carefully insert the index and middle fingers into the vaginal canal;
  * The participant will be instructed to contract the PFM in order to raise and compress the examiner's fingers.
  * To conclude, the participant will be directed to completely relax the PFM.

SECONDARY OUTCOMES:
International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) | 20 minutes
  Reports of urinary incontinence (UI) will be evaluated through the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF)at baseline and after 10 weeks. This questionnaire was translated and validated into the Portuguese language by Tamanini et al. (2004), and evaluates the symptoms, severity of UI, and the impact that UI has on women's quality of life (QoL). It is a brief questionnaire and the purpose of its use is to facilitate the comparison of data from different studies and to enable a more consistent and unified assessment of UI symptoms and its repercussion in QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Cristine HJ Ferreira, PhD, Principal Investigator — Ribeirão Preto Medical School, University of São Paulo
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ignacio Antonio F, Bo K, Pena CC, Bueno SM, Mateus-Vasconcelos ECL, Fernandes ACNL, Ferreira CHJ. Intravaginal electrical stimulation increases voluntarily pelvic floor muscle contractions in women who are unable to voluntarily contract their pelvic floor muscles: a randomised trial. J Physiother. 2022 Jan;68(1):37-42. doi: 10.1016/j.jphys.2021.12.004. Epub 2021 Dec 21. PMID 34952812